CLINICAL TRIAL: NCT06781775
Title: Gestational Diabetes Treatment: Should We Continue Metformin When Starting Insulin? a Randomized Control Trial
Brief Title: GDM: Insulin with or Without Metformin?
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christopher S. Ennen, Associate Professor, Division of Maternal Fetal Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 231576
Record Dates: First submitted 2024-03-18; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin; Insulin

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin + Insulin (Active Comparator): Pregnant women with gestational diabetes who have uncontrolled blood sugar on metformin alone will be started on insulin and will stay on metformin.
  Interventions: Drug: Metformin + Insulin
- Insulin (Active Comparator): Pregnant women with gestational diabetes who have uncontrolled blood sugar on metformin along will be started on insulin and metformin will be discontinued.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin + Insulin — Pregnant women who have have gestational diabetes and have uncontrolled blood sugar with metformin alone will stay on metformin and add insulin.
  Arms: Metformin + Insulin
Drug: Insulin — Pregnant women who have have gestational diabetes and have uncontrolled blood sugar with metformin alone will stop on metformin and add insulin.
  Arms: Insulin

SUMMARY:
This will be a randomized trial of patients with gestational diabetes who start hypoglycemic therapy with metformin but eventually require insulin. It will examine whether continuing metformin when adding insulin versus discontinuing metformin when insulin is added is beneficial. The investigators hypothesize that continuing metformin will reduce the needed insulin dosage and improve maternal and neonatal outcomes in these patients.

DETAILED DESCRIPTION:
This research study is being conducted to better treat patients who develop gestational diabetes which is diabetes that is diagnosed and present only during the course of pregnancy. Normally patients that develop gestational diabetes are treated with either metformin or insulin. Some need treatment with both. Both are considered safe in pregnancy and both are considered as standard treatments by national guidelines. Many patients ask to start with metformin because it is easy to take and does not require an injection. Sometimes, patients' blood sugars are not controlled enough on metformin so they need insulin to assist with control of the blood sugars. The investigators are studying patients who have tried metformin for gestational diabetes but did not have enough blood sugar control on metformin alone so they require insulin. The investigators are specifically looking at whether metformin should be continued when insulin is added or if metformin should be stopped. This has not been studied and nobody knows the correct answer on whether people should keep taking metformin when they need insulin or if they should stop the metformin. Some physicians decide to continue metformin with insulin and some do not since the investigators do not have an answer based on available research.

Patients will be split into two groups that are random. One group will continue metformin in addition to insulin and another group will stop taking metformin when insulin is needed to control their gestational diabetes. Some people may not want to take a pill and a shot and some may want to take a pill if it means taking less medication through shots.

This research questions is important because it will tell us how to better treat gestational diabetes and whether continuing metformin allows us to use less insulin. This could possibly mean less cost for the patient, a better medication schedule (less dose and/or less shots), better blood sugar control, better health benefits for the patient, and/or better health benefits for the baby.

This study is very similar to how current medical practice in obstetrics is currently as some providers continue metformin when insulin is needed and some discontinue it.

This research has not been done in patients with gestational diabetes before in this way. Metformin and insulin have been researched in pregnancy and are both considered standard treatments for gestational diabetes but they have not been researched like this together.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Pregnant female meeting diagnosis for gestational diabetes requiring medical treatment
4. Ability to take oral medication and be willing to adhere to the metformin regimen
5. Willing to take insulin if needed
6. Willing to take blood sugars 4 times per day

   -

   Exclusion Criteria:
   * 1) Metformin allergy or known intolerance, known hypersensitivity to insulin 2) Severe hepatic dysfunction 3) Chronic kidney disease 4) Pregnancy with major fetal anomalies 5) Non-viable pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
To determine if metformin reduces amount of insulin in patients with gestational diabetes who already require insulin | From enrollment into study until delivery, maximum 20 weeks
  Insulin dosage (units per kilogram body weight) at last visit prenatal visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No